CLINICAL TRIAL: NCT06429371
Title: Biopsychosocial Contributors to Irritability in Individuals With Shoulder Pain
Status: Recruiting | Type: Observational
Sponsor: University of Central Florida (Other)
Collaborators: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: 8
Record Dates: First submitted 2024-04-29; First posted 2024-05-28 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-05

CONDITIONS: Shoulder Pain
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individuals with Shoulder Pain: Individuals with shoulder pain that is at least 3/10 within the past 24 hours.
  Interventions: Other: Quantitative Sensory Testing; Other: Pain-Related Psychological Factors

INTERVENTIONS:
Other: Quantitative Sensory Testing — Participants will undergo heat pain threshold, cold pain threshold, pressure pain threshold, temporal summation, and conditioned pain modulation to characterize pain sensitivity.
Other: Pain-Related Psychological Factors — Participants will complete psychological questionnaires to characterize these factors.

SUMMARY:
Irritability was defined by Geoffrey Maitland as the vigor of activity to provoke symptoms, the severity of symptoms, and time for symptoms to subside. Irritability is deeply embedded in the physical therapy clinical decision-making process. However, the mechanisms contributing to irritability are unknown. Therefore, the purpose of this study is to characterize pain sensitivity and pain-related psychological factors by irritability level in individuals with shoulder pain.

ELIGIBILITY:
Inclusion Criteria:

* shoulder pain symptom intensity rated as 3/10 or higher in the past 24 hours
* attending physical therapy for shoulder pain

Exclusion Criteria:

* non-English speaking
* systemic medical conditions that affect sensation, such as uncontrolled diabetes
* history of shoulder surgery or fracture within the past 6 months
* history of a chronic pain condition, such as fibromyalgia
* blood clotting disorder, such as hemophilia
* contraindication to the application of ice (blood pressure > 140/90 mmHg, cold urticaria, cryoglobulinemia, paroxysmal cold hemoglobinuria, circulatory compromise)
* currently pregnant

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Individuals with shoulder pain
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-05-24 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Heat pain Threshold | Day 1
  A thermode will be applied to the deltoid, tibialis anterior, and lower back. The thermode will gradually increase temperature until the sensation changes from comfortable warmth to pain (pain threshold). Once pain threshold is reached, the temperature in degrees Celsius for heat pain threshold is recorded.
Cold Pain Threshold | Day 1
  A thermode will be applied to the deltoid, tibialis anterior, and lower back. The thermode will gradually decrease temperature until the sensation changes from comfortable cold to pain (pain threshold). Once pain threshold is reached, the temperature in degrees Celsius for cold pain threshold is recorded.
Pressure Pain Threshold | Day 1
  An algometer will be applied to the deltoid, tibialis anterior, and lower back. Pressure will be gradually applied until the sensation changes from comfortable pressure to pain (pain threshold). Once pain threshold is reached, the pressure in kilopascals will be recorded for pressure pain threshold.

CONTACTS AND LOCATIONS:
Overall Officials: Abigail Anderson, Principal Investigator — University of Central Florida
Locations (1):
- University of Central Florida, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided